CLINICAL TRIAL: NCT00043823
Title: Safety and Efficacy of Recombinant Humanized Monoclonal Anti-VEGF Antibody rhuMAb VEGF and EGFR Tyrosine Kinase Inhibitor OSI-774 for Locally Advanced or Metastatic Non-Squamous Cell NSCLC in Patients Who Have Been Previously Treated
Brief Title: Avastin and Tarceva for Locally Advanced or Metastatic Non-Squamous Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-604; VICC THO 0206
Record Dates: First submitted 2002-08-14; First posted 2002-08-15 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Lung Cancer; Avastin; Bevacizumab; rhuMAb VEGF; Anti-VEGF monoclonal antibody; Tarceva; OSI-774; Erlotinib Hydrocholoride
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avastin + Tarceva (Experimental): Combination Therapy (Avastin + Tarceva) = Avastin IV Day 1 of each 21-day cycle + oral Tarceva daily.
  Interventions: Drug: Avastin; Drug: Tarceva

INTERVENTIONS:
Drug: Avastin — 7.5 mg/kg By Vein on Day 1 of Every 21 Day Cycle
  Other Names: rhuMAb VEGF; Bevacizumab; Anti-VEGF monoclonal antibody
Drug: Tarceva — 100 mg By Mouth Daily for 3 Weeks
  Other Names: OSI-774; Erlotinib Hydrocholoride

SUMMARY:
Primary Objectives:

1. (Phase I) To establish the maximum tolerated dose and dose-limiting toxicities of the combination of OSI-774 (Tarceva™) and rhuMAb VEGF (Avastin™) in patients with advanced Non-small-cell lung carcinoma (NSCLC).
2. (Phase II) To assess response rate and tolerability of the regimen at the dose level established in the phase I portion of this study.

Secondary Objectives:

1. (Phase I and II) To evaluate the pharmacokinetic interaction between the combination.
2. (Phase I) To establish a phase II regimen of the OSI-774/ rhuMAb VEGF combination, for further study alone or in combination with cytotoxic chemotherapy.

DETAILED DESCRIPTION:
Patients will be treated with oral Tarceva daily for 21 days each cycle. Patients will receive Avastin by IV on day 1 of each 21-day cycle. If a patient has no grade 3 or 4 toxicities after the 1st cycle, then the patient may continue the same doses of Tarceva and Avastin for another cycle. If the patient has response or stable disease after 6 weeks (2 cycles), the patient may continue on the same doses of Tarceva and Avastin. A patient may receive treatment on this study for up to one year, unless his or her disease progresses or side effects become too severe.

The starting dose is 100 mg daily of Tarceva and 7.5 mg/kg every 21 days of Avastin.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically proven stage IIIB with pleural effusion, stage IV or recurrent non-squamous NSCLC.
* Patient has a Karnofsky performance status >=70%.
* Patient has adequate bone marrow function: WBC >= 3,000 cells/mm3, ANC >= 1,500 cells/mm3, platelet count >= 100,000 cells/mm3, Hgb >= 9.0 g/dL.
* Patient has adequate liver function: total bilirubin level <= 2.0 mg/dL, albumin >= 2.5 g/dL.
* Transaminases (aspartate aminotransferase (AST or SGOT) and/or alanine aminotransferase (ALT or SGPT)) and alkaline phosphatase may be up to 2.5 x ULN.
* Patient has adequate renal function: a serum creatinine < 2 mg/dl
* Patient has signed a written informed consent.
* Patient has received at least one prior chemotherapeutic regimen for recurrent or metastatic disease.

Exclusion Criteria:

* Patient has not received prior chemotherapeutic regimens for advanced disease.
* Patient has received prior biologic therapy targeting epidermal growth factor receptor (EGFR) and/or Vascular endothelial growth factor (VEGF).
* Patient has received radiation therapy within the past 3 weeks.
* Patient has signs or symptoms of acute infection requiring systemic therapy.
* Patient exhibits confusion, disorientation, or has a history of major psychiatric illness that may impair patient's understanding of the informed consent.
* Patient requires total parenteral nutrition with lipids.
* Patient has a history of uncontrolled heart disease and/or uncontrolled hypertension (> 150/100 mmHg).
* Because of the possible teratogenic effect, pregnant women and women who are currently breast-feeding may not participate in this study. - All women of childbearing potential must have a negative pregnancy test within 24 hours prior to enrolling in the study.
* Serious infection or other intercurrent illness requiring immediate therapy.
* Clinical/imaging evidence of Central Nervous System (CNS) malignancy or with recently treated CNS malignancy, as well as those experiencing recent cerebrovascular accident (CVA), or other CNS bleeding.
* Pediatric patients in whom open growth plates would be expected.
* Urine protein qualitative value of > 30 in urinalysis or > +1 in proteinuria testing by dipstick.
* Patient has a clinical history of coagulopathy or thrombosis.
* Patient is currently receiving or intending to receive anti-coagulants.
* Patient has had a recent myocardial infarction (still inside the healing period). Note: a six-month window is optimal.
* Patient is recovering from recent major surgery (e.g., less than 2 weeks since surgery) or is anticipating major surgery.
* Patient has a clinical history of hemoptysis or hematemesis.
* Patient may not have percutaneous endoscopic gastrostomy (PEG) or gastrostomy (G) tube.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2002-08-01 (Actual); Primary Completion 2006-05-15 (Actual); Study Completion 2006-05-15 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Tarceva in combination with Avastin | After each 21 day cycle

SECONDARY OUTCOMES:
Response in Patients With NSCLC Receiving Combination Avastin and Tarceva | 6 weeks (2 cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Roy S. Herbst, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org